CLINICAL TRIAL: NCT03612830
Title: Comparison of Laparoscopic and Endoscopic Cooperative Surgery and Robotic and Endoscopic Cooperative Surgery in the Operation of Gastric Submucosal Tumor
Brief Title: A Randomized Controlled Clinical Study on the Application of the Third Space in the Operation of Gastric Submucosal Tumor
Acronym: RECSINSMTs
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Collaborators: Air Force Military Medical University, China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: XJYFY-2018W411
Record Dates: First submitted 2018-04-13; First posted 2018-08-02 (Actual); Last update posted 2018-08-15 (Actual); Status verified 2018-04

CONDITIONS: Gastric Submucosal Tumors
Keywords: The Third Space

STUDY DESIGN:
Intervention Model Description: Laparoscopic and Endoscopic cooperative sugery,Robotic and Endoscopic cooperative sugery
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LECS (Experimental): Laparoscopic and Endoscopic cooperative surgery,LECS resects the tumor completely by laparoscopy with the help of the precise positioning and guidance of endoscopy .
  Interventions: Procedure: Laparoscopy endoscopy cooperated surgery
- RECS (Experimental): Robotic and Endoscopic cooperative surgery,RECS resects the tumor completely by Dan Vinchi robot with the help of the precise positioning and guidance of endoscopy .
  Interventions: Procedure: Dan Vinchi robot endoscopy cooperated surgery

INTERVENTIONS:
Procedure: Laparoscopy endoscopy cooperated surgery — LECS resects the tumor completely by laparoscopy with the help of the precise positioning and guidance of endoscopy
  Arms: LECS
Procedure: Dan Vinchi robot endoscopy cooperated surgery — RECS resects the tumor completely by Dan Vinchi Robot with the help of the precise positioning and guidance of endoscopy
  Arms: RECS

SUMMARY:
Gastric submucosal tumors (SMTs) are rare findings during routine upper endoscopy; the incidence of these lesions may be as high as 0.4%.SMTs display a wide spectrum,ranging from benign to highly malignant, with gastrointestinal stromal tumors (GISTs) being the most common type.SMTs is a gastrointestinal tumor,surgical operation is still the main method of gastric tumor treatment.The common surgical methods for resection of SMTs include laparotomy and laparoscopic surgery.In recent years, the Da Vinci robot assisted gastric resection has become a new way to treat gastric cancer. Compared with the traditional laparoscopy and laparotomy, the operation of the robot is more precise and flexible, with obvious advantages of minimally invasive and good application value and prospect.In recent years, some scholars have put forward the concept of the third space.The concept of the "third space" was initiatively proposed at the same time when new endoscopic surgery approach via natural orifice transluminal was put forward(NOTES). To be specific, with respect to the first space(lumen) and second space(peritoneal cavity),the third space refers to the intramural space.The aim of the study is to compare value (outcomes/costs) of surgery in patients with SMTs by 2 approaches:Laparoscopic and Endoscopic cooperative surgery(LECS),Robotic and Endoscopic cooperative surgery(RECS).First of all, the investigators will collect 80 cases of SMTs patients, randomly assigned for the LECS and RECS groups. Secondly, to analyzing the demographic data,basic treatment and follow-up data, including the operation time, blood loss, the number of cut edge positive, the distances of cut edge away from the tumor edge, average such confinement, the meal time, cost of treatment, tumor recurrence rate, the presence of residual stomach, upset stomach and frequency,complications and other indicators.

ELIGIBILITY:
Inclusion Criteria:

* Patients without contraindications gastroscope，surgery and anesthesia;
* Gastroscope found submucosal lesions, qualitative hard;Endoscopic ultrasonography (EUS) confirmed the lesions come from the muscularis propria;
* Tumors diameter > 2 cm;Or tumors had < 2 cm, but the position is located in the stomach wall, after nearly cardia and it is a difficult position for gastroscope ;
* Tumors diameter < 5 cm, the tumors had complete, no broken feed and bleeding;
* Not found the tumor metastasis;
* There is no history of abdominal surgery, no severe abdominal cavity adhesion
* Normal coagulation function;
* There is no history of anticoagulant drugs, or who take aspirin, salvia miltiorrhiza, etc., should stop taking drugs for more than one week;
* Patients and their families volunteered choice the surgical procedure and signed informed consent.

Exclusion Criteria:

* Patients with preoperative assessment of distant metastasis;
* Patients with preoperative radiation and chemotherapy or hormone therapy;
* Patients with acute obstruction, bleeding or perforation of the emergency surgery;
* Patients with a history of abdominal trauma or abdominal surgery;
* Patients with contraindications gastroscope，surgery and anesthesia.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-04-11 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
operation time | 1 hours to 6 hours through the surgery completion
  record in minutes,from the beginning of anesthesia to the end

SECONDARY OUTCOMES:
blood loss | 1 hours to 6 hours through the surgery completion
  from the surgical record sheet
success rate | from two days to two weeks after surgery
  to ensure the integrity of the tumor and obtain the negative surgical margin
time in bed | from two days to two weeks after surgery
  the time in bed to the postoperative patient
time to take food | from two days to two weeks after surgery
  the time to eat to the postoperative patient
postoperative complication rate | from two weeks to one year after surgery
  including anastomotic stoma fistula,anastomotic stenosis,abdominal infection,postoperative bleeding
tumor recurrence rate | from one month to 2 years after surgery
  periodic review the CT or MRI or endoscope
hospitalization expenses | 1 month
  total hospitalization expenses

CONTACTS AND LOCATIONS:
Overall Officials: Jun Jun She, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China